CLINICAL TRIAL: NCT07206342
Title: Evaluation of the Non-inferiority of Resorbable Gelatin Embolization Compared to Embolization Combined With Endometrial Aspiration for the Management of Hemorrhagic Uterine Vascular Abnormalities Following Premature Termination of Pregnancy
Acronym: NIEMBUT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Bordeaux (Other); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier Universitaire Saint Etienne, France, 43055 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38RC24.0406
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hemorrhage, Obstetric; Uterine Abnormality; Uterine Artery Embolization; Vaginal Bleeding During Pregnancy; Vaginal Bleeding
Keywords: abnormalities vascular uterine; embolization; intrauterine retention; hemorrhage; uterine artery embolization; vaginal bleedings; hysterectomy; uterine hemorrhage; embolization, therapeutic
MeSH Terms: conditions — Hemorrhage; Uterine Anomalies; Uterine Hemorrhage | interventions — Embolization, Therapeutic; ethylene-vinyl alcohol copolymer; Hysteroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the radiologist who performs the ultrasounds will be blinded to the evaluation of the primary judgment criterion (he will not have information regarding the group assigned to the patient).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- embolization therapy (Experimental): Patients will undergo embolization alone, which involves temporarily blocking the uterine artery or arteries supplying a hypervascular abnormality using resorbable gelatin fragments.
  Interventions: Procedure: embolization therapy
- Embolization followed by aspiration (Active Comparator): Patients will undergo embolization prior to endometrial aspiration. Embolization will be performed in the same manner as in group "Embolization alone" but will be followed within 48 hours by a second procedure to remove the intrauterine residue that will have been devascularized (= deprived of blood) by the embolization.
  Interventions: Procedure: embolization followed by aspiration

INTERVENTIONS:
Procedure: embolization therapy — Patients will undergo embolization alone, which involves temporarily blocking the uterine artery or arteries supplying a hypervascular abnormality using resorbable gelatin fragments.
  Other Names: embolic agent
  Arms: embolization therapy
Procedure: embolization followed by aspiration — Patients will undergo embolization prior to endometrial aspiration. Embolization will be performed in the same manner as in group "Embolization alone" but will be followed within 48 hours by a second procedure to remove the intrauterine residue that will have been devascularized (= deprived of blood) by the embolization.
  Other Names: endometrial aspiration; intrauterine aspiration; hysteroscopy
  Arms: Embolization followed by aspiration

SUMMARY:
The goal of this clinical trial is to determine the best treatment for patients who experience vaginal bleeding following a premature termination of pregnancy.

The main questions it aims to answer are:

* Evaluate the effectiveness of embolization alone versus embolization followed by aspiration in stopping bleeding
* Evaluate its effectiveness in restoring the menstrual cycle.
* What are the complications associated with the two procedures?
* What is their impact on future fertility?

The researchers will evaluate the patients over a period of 12 months.

Participants will:

* Undergo one of the two procedures (procedure 1: embolization alone and procedure 2: embolization combined with aspiration).
* Will participate in regular follow-ups to monitor the risk of recurrence of -bleeding and complications associated with the two treatments
* Will undergo imaging tests to assess the persistence of bleeding after the procedure

DETAILED DESCRIPTION:
Ten to 15% of pregnancies end in the first trimester. Voluntary termination of pregnancy and spontaneous miscarriage, the two main causes of pregnancy loss, are managed medically or surgically in order to remove the intrauterine residue and restore a vacant uterus. In cases of incomplete evacuation, uterine retention may persist in approximately 1% of all pregnancies and up to 40% of pregnancy terminations in the second trimester.

The management of uterine retention depends on the clinical presentation and its vascularization on ultrasound. If it is not vascularized or only slightly vascularized, simple aspiration or monitoring is considered. In cases of hypervascularity, treatment is debated given the variable amount of bleeding and the sometimes spontaneously favorable outcome. Doppler criteria (systolic peak velocity, resistance index, or vascular invasion of the myometrium) have been described to select patients who are likely to have a spontaneous favorable outcome from those who require invasive management. In cases of hypervascularized intrauterine retention with negative findings on Doppler ultrasound, performing endometrial aspiration carries a significant risk of severe bleeding during the procedure and is generally preceded by embolization in order to minimize this risk (embolization + aspiration). Aspiration induces adhesions (synechiae) that can impair the patient's future fertility.

Recent publications show the effectiveness of temporary embolization alone using resorbable gelatin fragments to stop bleeding. Our team has reported uterine emptiness rates of approximately 75% at 1 month and 95% at 3 months after embolization alone with resorbable gelatin.

The objective of this study is therefore to evaluate the non-inferiority of embolization alone with resorbable gelatin compared to embolization followed by endometrial aspiration in patients with hypervascularized and hemorrhagic intrauterine retention following premature termination of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Patient who experienced a miscarriage within 3 months
* Patient with gynecological bleeding
* Patient presenting with hypervascularized uterine retention with negative Doppler ultrasound findings (endometrial hypervascularization with 1) systolic peak velocity greater than 70 cm/s and/or 2) resistance index (RI) within the retention < 0.5)
* Patient affiliated to french social security
* Patient who has signed the written informed consent form

Exclusion Criteria:

* Patient presenting to the emergency department with hemorrhagic shock: systolic blood pressure < 90 mmHg associated with tachycardia > 120 bpm
* Severe renal failure (glomerular filtration rate < 30 mL/min)
* Medical history of severe allergy to iodinated contrast media
* Severe coagulation disorders (platelets <50G/L, PT < 50%)
* Anticoagulant and/or antiplatelet agent that cannot be discontinued a few days before the procedure
* Patient referred to in Articles L1121-5, L1121-6, and L1121-8 of the French Public Health Code
* Staff with a hierarchical relationship to the principal investigator
* Patient in the exclusion period of another study
* Patient cannot be contacted in an emergency
* Participation in other interventional studies during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical success post-procedure as assessed by Doppler-ultrasound | From baseline to 3 months after procedure
  The primary endpoint is clinical success defined by a null uterine cavity on follow-up Doppler ultrasound and no persistent or recurrent bleeding requiring a new procedure

SECONDARY OUTCOMES:
Persistence or recurrence of bleeding at 1 month follow-up in both groups. | From baseline to 1 month
  Evaluate the effectiveness of embolization alone versus embolization followed by aspiration at 1 month of follow-up in stopping bleeding in patients with hypervascularized hemorrhagic uterine retention following premature termination of pregnancy.
Safety of both treatments | Fom intervention to 90 days after
  Complications attributable to procedures within 90 days of admission according to the Clavien-Dindo classification
the effectiveness of embolization alone compared to embolization followed by uterine evacuation at 1 month after procedure | From intervention to 1 month
  Measurement of uterine emptiness on Doppler ultrasound at 1 month
the effectiveness of embolization alone compared to embolization followed by uterine evacuation at 3 months after procedure | From intervention to 3 months
  Measurement of uterine emptiness on Doppler ultrasound at 3 months
the impact of embolization alone compared to embolization followed by aspiration on the resumption of the menstrual cycle | From intervention to 12 months
  Time between intervention and resumption of menstrual cycle
the impact of embolization alone versus embolization followed by aspiration on subsequent fertility | From intervention to 12 months
  New pregnancy occurring within 12 months of the patient's admission
If infertility diagnosis within 12 months, the rate of synechiae found between the two groups. | From intervention to 12 months
  Uterine adhesions on hysteroscopy performed for infertility assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Ghelfi, Principal Investigator — CHU Grenoble Alpes
Locations (4):
- France (4):
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand-Gabriel Montpied, Clermont-Ferrand
  - CHU Grenoble Alpes, Grenoble
  - CHU de St Etienne-Hôpital Nord, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCracken G, Houston P, Lefebvre G; Society of Obstetricians and Gynecologists of Canada. Guideline for the management of postoperative nausea and vomiting. J Obstet Gynaecol Can. 2008 Jul;30(7):600-7, 608-16. doi: 10.1016/s1701-2163(16)32895-x. English, French. PMID 18644183
- [Background] Huchon C, Drioueche H, Koskas M, Agostini A, Bauville E, Bourdel N, Fernandez H, Fritel X, Graesslin O, Legendre G, Lucot JP, Panel P, Raiffort C, Giraudet G, Bussieres L, Fauconnier A. Operative Hysteroscopy vs Vacuum Aspiration for Incomplete Spontaneous Abortion: A Randomized Clinical Trial. JAMA. 2023 Apr 11;329(14):1197-1205. doi: 10.1001/jama.2023.3415. PMID 37039805
- [Background] Kimura Y, Osuga K, Nagai K, Hongyo H, Tanaka K, Ono Y, Higashihara H, Matsuzaki S, Endo M, Kimura T, Tomiyama N. The efficacy of uterine artery embolization with gelatin sponge for retained products of conception with bleeding and future pregnancy outcomes. CVIR Endovasc. 2020 Feb 12;3(1):13. doi: 10.1186/s42155-020-00107-4. PMID 32052234
- [Background] Mathieu E, Riethmuller D, Delouche A, Sicot M, Teyssier Y, Finas M, Guillaume B, Thony F, Ferretti G, Ghelfi J. Management of Symptomatic Vascularized Retained Products of Conception by Proximal Uterine Artery Embolization with Gelatin Sponge Torpedoes. J Vasc Interv Radiol. 2022 Nov;33(11):1313-1320. doi: 10.1016/j.jvir.2022.07.018. Epub 2022 Jul 19. PMID 35868595
- [Background] Deans R, Abbott J. Review of intrauterine adhesions. J Minim Invasive Gynecol. 2010 Sep-Oct;17(5):555-69. doi: 10.1016/j.jmig.2010.04.016. Epub 2010 Jul 24. PMID 20656564
- [Background] Tam WH, Lau WC, Cheung LP, Yuen PM, Chung TK. Intrauterine adhesions after conservative and surgical management of spontaneous abortion. J Am Assoc Gynecol Laparosc. 2002 May;9(2):182-5. doi: 10.1016/s1074-3804(05)60129-6. PMID 11960045
- [Background] Gilbert A, Thubert T, Dochez V, Riteau AS, Ducloyer M, Ragot P, Frampas E, Douane F, David A. Angiographic findings and outcomes after embolization of patients with suspected postabortion uterine arteriovenous fistula. J Gynecol Obstet Hum Reprod. 2021 Sep;50(7):102033. doi: 10.1016/j.jogoh.2020.102033. Epub 2020 Dec 7. PMID 33301980
- [Background] Camacho A, Ahn EH, Appel E, Boos J, Nguyen Q, Justaniah AI, Faintuch S, Ahmed M, Brook OR. Uterine Artery Embolization with Gelfoam for Acquired Symptomatic Uterine Arteriovenous Shunting. J Vasc Interv Radiol. 2019 Nov;30(11):1750-1758. doi: 10.1016/j.jvir.2019.04.002. Epub 2019 Aug 10. PMID 31409569
- [Background] Vyas S, Choi HH, Whetstone S, Jha P, Poder L, Shum DJ. Ultrasound features help identify patients who can undergo noninvasive management for suspected retained products of conception: a single institutional experience. Abdom Radiol (NY). 2021 Jun;46(6):2729-2739. doi: 10.1007/s00261-020-02948-y. Epub 2021 Jan 18. PMID 33459841
- [Background] Timmerman D, Wauters J, Van Calenbergh S, Van Schoubroeck D, Maleux G, Van Den Bosch T, Spitz B. Color Doppler imaging is a valuable tool for the diagnosis and management of uterine vascular malformations. Ultrasound Obstet Gynecol. 2003 Jun;21(6):570-7. doi: 10.1002/uog.159. PMID 12808674
- [Background] Kamaya A, Petrovitch I, Chen B, Frederick CE, Jeffrey RB. Retained products of conception: spectrum of color Doppler findings. J Ultrasound Med. 2009 Aug;28(8):1031-41. doi: 10.7863/jum.2009.28.8.1031. PMID 19643786
- [Background] Foreste V, Gallo A, Manzi A, Riccardi C, Carugno J, Sardo ADS. Hysteroscopy and Retained Products of Conception: An Update. Gynecol Minim Invasive Ther. 2021 Nov 5;10(4):203-209. doi: 10.4103/GMIT.GMIT_125_20. eCollection 2021 Oct-Dec. PMID 34909376
- [Background] Quenby S, Gallos ID, Dhillon-Smith RK, Podesek M, Stephenson MD, Fisher J, Brosens JJ, Brewin J, Ramhorst R, Lucas ES, McCoy RC, Anderson R, Daher S, Regan L, Al-Memar M, Bourne T, MacIntyre DA, Rai R, Christiansen OB, Sugiura-Ogasawara M, Odendaal J, Devall AJ, Bennett PR, Petrou S, Coomarasamy A. Miscarriage matters: the epidemiological, physical, psychological, and economic costs of early pregnancy loss. Lancet. 2021 May 1;397(10285):1658-1667. doi: 10.1016/S0140-6736(21)00682-6. Epub 2021 Apr 27. PMID 33915094